CLINICAL TRIAL: NCT06496568
Title: A Phase I/Ib Study Evaluating Single-Agent Inavolisib and Inavolisib Plus Atezolizumab in PIK3CA-Mutated Cancers
Brief Title: A Study Evaluating Single-agent Inavolisib and Inavolisib Plus Atezolizumab in PIK3CA-Mutated Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO43909; 2021-006618-36 (EudraCT Number)
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: PIK3CA-Mutated Cancers
MeSH Terms: interventions — inavolisib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants in this group will receive inavolisib tablets, to be taken by mouth (PO), once daily (QD), on Days 1-21 of each cycle.
  Interventions: Drug: Inavolisib
- Arm B (Experimental): Participants in this group will receive inavolisib tablets, to be taken PO, QD and atezolizumab given as an intravenous (IV) infusion once every 3 weeks (Q3W).
  Interventions: Drug: Inavolisib; Drug: Atezolizumab

INTERVENTIONS:
Drug: Inavolisib — Participants will receive inavolisib, 9 milligram (mg), PO, QD on Days 1-21 of each 21-day cycle.
Drug: Atezolizumab — Participants will receive atezolizumab, 1200 mg, as IV infusion Q3W on Day 1 of each 21-day cycle.
  Arms: Arm B

SUMMARY:
The purpose of the study is to assess the safety and efficacy of inavolisib as a single-agent and in combination with atezolizumab in participants with phosphatidylinositol 4,5-bisphosphate 3-kinase catalytic subunit alpha isoform (PIK3CA)-mutated cancers, including previously treated head and neck squamous cell carcinoma (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent and/or metastatic HNSCC that has been previously treated with systemic therapy in the recurrent and/or metastatic setting
* Documented positive or negative human papillomavirus (HPV) status as determined locally by p16 immunohistochemistry (IHC; preferred), in situ hybridization, and/or by polymerase chain reaction-based assay
* Eligible participants must not be suitable for treatment with surgery and/or radiation
* Confirmation of biomarker eligibility: Valid results from either central testing of blood or local testing of blood or tumour tissue documenting PIK3CA-mutated tumour status
* Consent to provide fresh (preferred) or archival tumour tissue specimen
* Negative hepatitis B surface antigen (HBsAg) and total hepatitis B core antibody (HBcAb) test or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* Measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of >=12 weeks

Exclusion Criteria:

* Prior treatment with any phosphatidylinositol 3-kinase (PI3K), protein kinase B (AKT), or mammalian target of rapamycin (mTOR) inhibitor, or any agent whose mechanism of action is to inhibit the PI3K/AKT/mTOR pathway
* Appropriate for treatment with surgery and/or radiation at the time of entry into the study, as per national or local treatment guidelines
* Type II diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type I diabetes
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Known and untreated, or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Participants with a history of treated CNS metastases are eligible provided they meet specified criteria
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures twice per week or more frequently
* Serious infection requiring IV antibiotics within 7 days prior to Day 1 of Cycle 1
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of the need for such a vaccine during study treatment
* Any concurrent ocular or intraocular condition (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, would require medical or surgical intervention during the study period to prevent or treat vision loss that might result from that condition
* Active inflammatory (e.g., uveitis or vitritis) or infectious (e.g., conjunctivitis, keratitis, scleritis, or endophthalmitis) conditions in either eye or history of idiopathic or autoimmune-associated uveitis in either eye
* Requirement for daily supplemental oxygen
* Symptomatic active lung disease, including pneumonitis
* History of or active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis) or any active bowel inflammation (including diverticulitis)
* Known Human Immunodeficiency Virus (HIV) infection
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, metabolic, or infectious disease) or any other diseases, active or uncontrolled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or that renders the participant at high risk from treatment complications
* Chemotherapy, radiotherapy, or any other anti-cancer therapy within 2 weeks before enrolment
* Investigational drug(s) within 4 weeks before enrolment
* Unresolved toxicity from prior therapy, except for hot flashes, alopecia, and Grade <=2 peripheral neuropathy
* History of other malignancy within 5 years prior to screening, with specified exceptions
* History of or active clinically significant cardiovascular dysfunction
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study)
* Chronic corticosteroid therapy of >=10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressants for a chronic disease
* Allergy or hypersensitivity to components of the inavolisib formulation
* Treatment with strong CYP3A4 inducers or strong CYP3A4 inhibitors within 1 week or five drug-elimination half-lives, whichever is longer, prior to initiation of study treatment
* Major surgical procedure, or significant traumatic injury, within 28 days prior to Day 1 of Cycle 1; or anticipation of the need for major surgery during study treatment
* Minor surgical procedures <7 days prior to the first dose of study treatment

Exclusion criteria specific to arms utilizing atezolizumab:

* Prior serious immune-mediated toxicities resulting from treatment with any checkpoint inhibitor including, but not limited to, atezolizumab, pembrolizumab, or nivolumab
* Treatment with any checkpoint inhibitor within 5 half-lives of Day 1 of Cycle 1
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with specified exceptions
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan; a history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteraemia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment; participants receiving prophylactic antibiotics may be eligible for the study
* Prior allogeneic stem cell or solid organ transplantation
* Current treatment with anti-viral therapy for HBV
* Treatment with systemic immunostimulatory agents within 4 weeks or five drug-elimination half-lives of the drug (whichever is longer)
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of the need for systemic immunosuppressive medication during study treatment, with specified exceptions
* Poor peripheral venous access that would preclude repeated IV infusions
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Select Treatment-related Toxicities (TRT) in Arm B | Day 1 of Cycle 1 to Day 3 of Cycle 2 (each cycle = 21 days)
Percentage of Participants with Adverse Events (AEs) and serious adverse events (SAEs) | From baseline up to approximately 3 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Every 9 weeks from Day 1 of Cycle 1 during the first 2 years, and every 12 weeks thereafter until disease progression or initiation of another anti-cancer therapy whichever occurs first (up to approximately 3 years)
Best Objective Response (BOR) | Every 9 weeks from Day 1 of Cycle 1 during the first 2 years, and every 12 weeks thereafter until disease progression or initiation of another anti-cancer therapy whichever occurs first (up to approximately 3 years)
Duration of Response (DOR) | Every 9 weeks from Day 1 of Cycle 1 during the first 2 years, and every 12 weeks thereafter until disease progression or initiation of another anti-cancer therapy whichever occurs first (up to approximately 3 years)
Clinical Benefit Rate (CBR) | Every 9 weeks from Day 1 of Cycle 1 during the first 2 years, and every 12 weeks thereafter until disease progression or initiation of another anti-cancer therapy whichever occurs first (up to approximately 3 years)
Progression-free Survival (PFS) | Every 9 weeks from Day 1 of Cycle 1 during the first 2 years, and every 12 weeks thereafter until disease progression or initiation of another anti-cancer therapy whichever occurs first (up to approximately 3 years)
Plasma Concentration of Inavolisib in Arm A | Predose and 3 hours post-dose on Day 1 of Cycle 1 and 2 and at predose on Day 1 of Cycle 3 (each cycle = 21 days)
Area Under the Concentration-time Curve (AUC) of Inavolisib in Arm A | Predose and 3 hours post-dose on Day 1 of Cycle 1 and 2 and at predose on Day 1 of Cycle 3 (each cycle = 21 days)
Maximum Plasma Concentration (Cmax) of Inavolisib in Arm A | Predose and 3 hours post-dose on Day 1 of Cycle 1 and 2 and at predose on Day 1 of Cycle 3 (each cycle = 21 days)
Minimum Plasma Concentration (Cmin) of Inavolisib in Arm A | Predose and 3 hours post-dose on Day 1 of Cycle 1 and 2 and at predose on Day 1 of Cycle 3 (each cycle = 21 days)
Plasma Concentration of Inavolisib in Arm B | Predose and 3 hours post-dose on Day 1 of Cycle 1 and 2 and Predose on Day 1 of Cycle 3 (each cycle = 21 days)
AUC of Inavolisib in Arm B | Predose and 3 hours post-dose on Day 1 of Cycle 1 and 2 and Predose on Day 1 of Cycle 3 (each cycle = 21 days)
Cmax of Inavolisib in Arm B | Predose and 3 hours post-dose on Day 1 of Cycle 1 and 2 and Predose on Day 1 of Cycle 3 (each cycle = 21 days)
Cmin of Inavolisib in Arm B | Predose and 3 hours post-dose on Day 1 of Cycle 1 and 2 and Predose on Day 1 of Cycle 3 (each cycle = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (3):
  - Moores Cancer Center at UC San Diego Health, La Jolla, California
  - California Cancer Associates for Research & Excellence, Inc., San Marcos, California
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
- Canada (3):
  - BC Cancer Vancouver Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No